CLINICAL TRIAL: NCT05364333
Title: Effect of Remote Ischemic Preconditioning on Acute Kidney Injury in Patients Undergoing Heart Transplantation
Brief Title: Remote Ischemic Preconditioning and Acute Kidney Injury in HTX
Acronym: RIPCAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-1240
Record Dates: First submitted 2022-05-04; First posted 2022-05-06 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Heart Transplantation
Keywords: orthotopic heart transplantation; HTX

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham RIPC (Sham Comparator): Control patients will be submitted to 3 cycles of sham RIPC. Each cycle of Sham RIPC consists of a pseudo ischemia of the left upper limb caused by inflating a blood pressure cuff to 20mmHg for 5 minutes followed by 5 minutes of reperfusion time.
  Interventions: Procedure: Remote ischemic preconditioning
- RIPC (Experimental): Patients in the intervention group will be submitted to 3 cycles of RIPC. For each cycle of RIPC, a blood pressure cuff will be inflated at 200mmHg for 5 minutes (or at least 50mmHg above the systolic arterial blood pressure) followed by 5 minutes of reperfusion time.
  Interventions: Procedure: Remote ischemic preconditioning

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — For each cycle of RIPC, a blood pressure cuff will be inflated to the non-dominant arm at 200mmHg for 5 minutes (or at least 50mmHg above the systolic arterial blood pressure) followed by 5 minutes of reperfusion time

SUMMARY:
Postoperative Acute Kidney Injury (AKI) is a common complication after heart transplantation (HTX) affecting outcome of patients. Remote ischemic preconditioning (RIPC) is an intervention that showed positive effect on incidence of AKI in elective cardiac surgery. Effects of RIPC on AKI in HTX patients have not been investigated to date. Recently new biomarkers have been established, showing high sensitivity and specificity for AKI. Especially, Insulin-Like Growth Factor Binding Protein 7 (IGFBP7) together with Tissue Inhibitor of Metalloproteinases-2 (TIMP-2), known as nephrocheck®, are diagnostic biomarkers in this context. Hence, the investigators want to conduct a randomized controlled feasibility and proof of concept trial to determine the effects of RIPC on AKI after HTX, defined/detected using postoperative urinary [TIMP-2]*[IGFBP-7] concentration.

DETAILED DESCRIPTION:
Postoperative Acute Kidney Injury (AKI) is a common complication after heart transplantation (HTX) affecting outcome of patients. Anesthesia- and surgery-related factors, but also hemodynamic instability and nephrotoxic drugs are triggering AKI and are frequent in HTX patients. A recent meta-analysis showed that incidences of AKI (according to KDIGO criteria) and AKI requiring renal replacement therapy (RRT) after HTX are 62.8% and 11.8% respectively. Crucially, AKI post HTX is associated with reduced short term and 1-year patient survival as well as long-term outcome. Impaired baseline renal function due to heart failure is a main risk factor for AKI in patients undergoing heart transplant surgery. Our recent data shows that postoperative AKI requiring RRT is also frequent in patients with adequate baseline renal function after HTX. Again, nephrotoxicity of immunosuppressive drugs and treatment of hemodynamic instability by vasopressors showed relevance in risk prediction of AKI. Due to the high incidence of AKI and its strong effect on patient outcome and with regard to the increasing cases of end stage heart failure and Heart transplant surgery in recent years, AKI prevention holds promise to relevant outcome improvement in the future. However, recommended interventions to prevent AKI, i.e. avoidance of nephrotoxic drugs, improvement of hemodynamics or fluid therapy are limited in this specific setting. Thus, it is of big interest to identify procedures which could reduce AKI after HTX.

Remote ischemic preconditioning (RIPC) has been suggested in this context and the effects of RIPC on AKI have been investigated by several studies in the cardiac surgery setting. RIPC achieves ischemic preconditioning by non-invasive repetitive induction of limb ischemia blood pressure cuff. Thus, it is an intervention with barely relevant adverse effects. Moreover, RIPC is an investigator-independent and cost-effective procedure.

Zarbock et al. showed in a randomized clinical trial (RCT) that RIPC compared with no RIPC significantly reduced the rate of AKI and use of RRT in 240 patients undergoing on-pump coronary artery bypass graft (CABG) or valvular surgery. Although these results could be replicated by another single center RIPC trial, other RCTs could not show effects of RIPC on AKI. However, a recent meta-analysis of randomized controlled trials shows favorable effects of RIPC on incidence of AKI in patients undergoing cardiac surgery. Referring to the lack of alternatives, the high incidence of AKI and its deleterious long-term sequelae, RIPC is worth to be investigated as a promising strategy for renal protection after HTX. Of note, previous results from studies in the CABG or valvular surgery setting cannot be translated to patients undergoing HTX. Although cardiopulmonary bypass (CPB) is used in all of these patients, the hemodynamic situation after CPB can be different in patients with or without HTX when extracorporeal life support systems are used.

Recently new biomarkers have been established, showing high sensitivity and specificity for AKI. Especially, Insulin-Like Growth Factor Binding Protein 7 (IGFBP7) together with Tissue Inhibitor of Metalloproteinases-2 (TIMP-2), known as nephrocheck®, are diagnostic biomarkers in this context. Both intracellular proteins are released during tubular epithelial stress, as present during AKI. Those markers may help to better understand the effects of RIPC on AKI.

To date there are no RCTs investigating the effects of RIPC on postoperative AKI in this specific population of HTX patients. Hence, the investigators want to conduct a randomized controlled feasibility and proof of concept trial to determine the effects of RIPC on AKI after HTX, defined/detected using urinary [TIMP-2]*[IGFBP-7] concentration. Moreover, the investigators will analyze the impact of RIPC on renal and cardiac function as well as other important clinical outcomes as secondary endpoints. If this feasibility and proof-of-concept trial will have a positive result in terms of 1) the effect of the intervention and 2) the feasibility of our study design, the investigators will conduct a pragmatic multicenter RCT to answer the question if RIPC can really improve outcome of patients undergoing HTX.

ELIGIBILITY:
Inclusion Criteria:

- adult patients (>18 years) undergoing HTX

Exclusion Criteria:

* Acute myocardial infarction up to 7 days before surgery
* age younger than 18 years
* pre-existing AKI
* previous kidney transplantation
* chronic kidney disease with a glomerular filtration rate less than 30ml/min
* pregnancy
* peripheral vascular disease affecting the upper limbs
* hepato-renal syndrome
* drug therapy with sulfonamide or nicorandil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
postoperative TIMP2-IGFBP7 concentration | first 48 hours after HTX (arrival ICU, 24 hours after HTX, 48 hours after HTX)
  change in postoperative TIMP2-IGFBP7 concentration measured in urine of patients

SECONDARY OUTCOMES:
Postoperative urinary biomarker concentration | first 48 hours after HTX (arrival ICU, 24 hours after HTX, 48 hours after HTX)
  change in postoperative biomarker (NGAL, KIM-1, DKK3) concentration
AKI and renal replacement therapy | first 72 hours
  early AKI or need for renalreplacement therapy
Major adverse kidney events (MAKE) | during 30 days after HTX
  MAKE = death, renal replacement therapy, worsened kidney function
Major adverse cardiovascular events (MACE) | during 30 days after HTX
  MACE = cardiac death, stroke, non fatal myocardial infarction, new arrhythmia, deterioration due to congestive heart failure
Days alive and out of hospital | during 30 days after HTX
  days spent alive and out of the hospital

CONTACTS AND LOCATIONS:
Overall Officials: René M'Pembele, M.D., Principal Investigator — Heinrich-Heine University, Duesseldorf
Locations (1):
- University Hospital Duesseldorf, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No